CLINICAL TRIAL: NCT02492100
Title: A Multimodal Intervention to Address Sexual Dysfunction in Hematopoietic Stem Cell Transplant Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, El-Jawahri, Areej,M.D., Principal Investigator, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 15-158
Record Dates: First submitted 2015-07-02; First posted 2015-07-08 (Estimated); Results first posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: Sexual Dysfunction
Keywords: Sexual Dysfunction Post-Bone Marrow Transplant
MeSH Terms: conditions — Sexual Dysfunction, Physiological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Multi-modality sexual dysfunction intervention (Experimental): - Patients in remission > 6 months after allogeneic bone marrow transplant
  * Patient Enrollment and Baseline Data Collection
  * First Intervention Visit:
    * Comprehensive assessment of sexual dysfunction
    * Normalization & Education
    * Therapeutic interventions
    * Referral to Sexual Health Clinic if applicable
  * Follow-Up Intervention Visit --- Referral to Sexual Health Clinic if applicable
  Interventions: Behavioral: Multi-modality sexual dysfunction intervention

INTERVENTIONS:
Behavioral: Multi-modality sexual dysfunction intervention

SUMMARY:
This research study is evaluating the feasibility and impact of an intervention to improve sexual function in stem cell transplant survivors on participants' sexual function, quality of life, and mood.

- It is expected that about 50 stem cell transplant survivors will take part in this research study.

DETAILED DESCRIPTION:
Frequently survivors of stem cell transplantation report significant problems with their sexual function that impacts their quality of life, mood, and their intimacy and relationship with their partners. These issues can be very distressing to patients and their loved ones. The study doctors want to know if the introduction of an intervention focused on improving sexual function may improve a participant's overall care and quality of life.

The intervention includes a comprehensive assessment by a transplant clinician who is trained in sexual dysfunction assessment to explore the reasons for sexual dysfunction and focus on ways to improve the participant's symptoms. The study will use a series of questionnaires to measure a participant's sexual function, quality of life, and mood.

The main purpose of this study is examine whether this intervention is feasible and helpful for participants in terms of improving their symptoms and overall quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years) with hematologic malignancy who underwent an allogeneic HCT at least 6 months prior to study enrollment.
* Ability to speak English or able to complete questionnaires with assistance required from an interpreter or family member.
* Positive screen for sexual dysfunction that is causing distress based on the National Comprehensive Cancer Network survivorship guidelines

Exclusion Criteria:

* Patients with relapsed disease post-HCT.
* Significant psychiatric or other co-morbid disease, which the treating clinician believes prohibits the patient's ability to participate in the informed consent procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2015-06; Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Areej El-Jawahri, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm Pre and Post Sexual Health Intervention: A total of 47 patients who screened positive for sexual dysfunction causing distress agreed to participate in this pre-/post- design single-arm study
Period: Overall Study
Arm/Group | Single Arm Pre and Post Sexual Health Intervention
Started | 47
Completed | 46
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Groups:
- Multi-modality Sexual Dysfunction Intervention: - Patients in remission > 6 months after allogeneic bone marrow transplant
  * Patient Enrollment and Baseline Data Collection
  * First Intervention Visit:
    * Comprehensive assessment of sexual dysfunction
    * Normalization & Education
    * Therapeutic interventions
    * Referral to Sexual Health Clinic if applicable
  * Follow-Up Intervention Visit --- Referral to Sexual Health Clinic if applicable
  Multi-modality sexual dysfunction intervention
Arm/Group | Multi-modality Sexual Dysfunction Intervention
Number analyzed (Participants) | 47
Age, Continuous [Median (Full Range); unit: years] | 52.5 [24 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 44
  More than one race | 1
  Unknown or Not Reported | 0
Global satisfaction with sex [Mean (Standard Deviation); unit: units on a scale] — score ranges from 3-20 with higher scores indicating more satisfaction
  units on a scale | 16.07 (8.16)
Interest in sex [Mean (Standard Deviation); unit: units on a scale] — raw score ranges from 2-20 with higher scores indicating more interest in sex
  units on a scale | 10.98 (3.88)
quality of life [Mean (Standard Deviation); unit: units on a scale] — quality of life measured by FACT-BMT with score range of 0-164 with higher score indicating better quality of life
  units on a scale | 107.98 (22.00)
Depression (HADS) [Mean (Standard Deviation); unit: units on a scale] — using the HADS-Depression, score range 0-21 with higher score indicating higher depression symptoms.
  units on a scale | 4.28 (3.10)
Anxiety (HADS) [Mean (Standard Deviation); unit: units on a scale] — using the HADS-Anxiety score range 0-21, with higher scores indicating higher anxiety symptoms.
  units on a scale | 4.59 (3.32)

OUTCOME MEASURES:

1. Primary Outcome: Feasibility Primary Endpoint
Description: intervention deemed feasible if at least 75% of patients screening positive for sexual dysfunction causing distress agree to participate and at least 80% complete at least one additional follow-up visit. This is not a composite outcome. Study is deemed feasible (yes) if both criteria are met.
Time Frame: 6 months
Population: overall 94% (47 of 50) patients who screened positive for sexual dysfunction agreed to participate in the study and 80% attended at least 2 intervention visits
Measure: Count of Participants; unit: Participants
Groups:
- Single Arm Study: single arm study, pre/post design
Arm/Group | Single Arm Study
Number analyzed (Participants) | 47
Participants | 38

2. Secondary Outcome: Change in Sexual Function: Promis Sexual Function and Satisfaction Measure
Description: Interest in sex at 6 months, raw score range 2-20 with higher scores indicating higher interest.
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Singe Arm Pre/Post Design: single arm pre/post design
Arm/Group | Singe Arm Pre/Post Design
Number analyzed (Participants) | 46
units on a scale | 15.39 (3.69)

3. Secondary Outcome: Change in Quality of Life: Functional Assessment of Cancer Therapy- Bone Marrow Transplant
Description: quality of life at 6 months compared to baseline using the Functional Assessment of Cancer Therapy - Bone Marrow Transplant. Score range 0-164 with higher score indicating better quality of life.
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Singe Arm Pre/Post Design
Number analyzed (Participants) | 46
units on a scale | 123.88 (17.10)

4. Secondary Outcome: Change in Psychological Distress Scores - Hospital and Anxiety Depression Scale and Patient Health Questionnaire-9
Description: change in HADS depression score, depression subscale of the HADS has a score range of 0-21, with higher scores indicating more depression symptoms.
Time Frame: Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Single Arm Study
Number analyzed (Participants) | 46
units on a scale | 2.33 (2.56)

ADVERSE EVENTS:
Time Frame: 6 months
Description: no adverse events
Arm/Group | Single Arm Study
All-Cause Mortality (participants affected / at risk) | 1/47
Serious Adverse Events (participants affected / at risk) | 0/47
Other Adverse Events (participants affected / at risk) | 0/47

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-28): https://cdn.clinicaltrials.gov/large-docs/00/NCT02492100/Prot_SAP_000.pdf